CLINICAL TRIAL: NCT00479557
Title: A Phase Iia, Multicenter, Randomized, Third-party Unblinded, Adjuvant And Placebo-controlled, Multiple Ascending Dose, Safety, Tolerability And Immunogenicity Trial Of Acc-001 And Qs-21 Adjuvant In Subjects With Mild To Moderate Alzheimer's Disease
Brief Title: Study Evaluating Safety, Tolerability, And Immunogenicity Of ACC-001 In Subjects With Mild To Moderate Alzheimer's Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Collaborators: Janssen Alzheimer Immunotherapy (JAI) Research and Development, LLC (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 3134K1-200; B2571004 (Other: Alias Study Number); 2006-002061-39 (EudraCT Number)
Record Dates: First submitted 2007-05-24; First posted 2007-05-28 (Estimated); Results first posted 2016-01-01 (Estimated); Last update posted 2016-01-01 (Estimated); Status verified 2015-11

CONDITIONS: Alzheimer Disease
Keywords: Alzheimer's Disease; active immunization
MeSH Terms: conditions — Alzheimer Disease | interventions — vanutide cridificar; saponin QA-21V1

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 1 (Active Comparator): arm 1: ACC-001 (Vanutide Cridificar)+ QS-21
  Interventions: Biological: ACC-001 + QS-21
- 2 (Active Comparator): arm 2: ACC-001
  Interventions: Biological: ACC-001
- 3 (Placebo Comparator): arm 3: QS-21
  Interventions: Biological: QS-21
- 4 (Placebo Comparator): Drug: Phosphate Buffered Saline (PBS)
  Interventions: Drug: Placebo: Phosphate buffered saline

INTERVENTIONS:
Biological: ACC-001 + QS-21 — Vanutide Cridificar (3, 10, 30µg) + QS-21 (50µg), IM on day 1, month 1, month 3, month 6 and month 12
  Arms: 1
Biological: ACC-001 — Vanutide Cridificar (10, 30µg), IM on day 1, month 1, month 3, month 6 and month 12
  Arms: 2
Biological: QS-21 — QS-21 (50µg), IM on day 1, month 1, month 3, month 6 and month 12
  Arms: 3
Drug: Placebo: Phosphate buffered saline — Phosphate buffered Saline (pH : 7.4), IM on day 1, month 1, month 3, month 6 and month 12
  Arms: 4

SUMMARY:
To assess the safety, tolerability, and immunogenicity of ACC-001, an investigational active immunization, in patients with mild to moderate Alzheimer's disease.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of probable Alzheimer's Disease with Mini-Mental State Examination (MMSE) score of 16-26 (except Germany: 21-26)
* Brain MRI consistent with Alzheimer Disease
* Concurent use of Chloniesterase inhibitor or memantine allowed if stable
* Other inclusion criteria apply

Exclusion Criteria:

* Significant Neurological Disease other than Alzheimer's disease
* Major psychiatric disorder
* Contraindication to undergo brain MRI
* Clinically significant systemic illness
* Other exclusion criteria apply

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2007-05; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (23):
- France (12):
  - Groupe Hospitalier Pitie-Salpetriere, Paris, Cedex 13 (mri)
  - Hôpital Pitié-Salpétrière, Paris, Paris
  - Hopital Pellegrin-Centre Mémoire de Recherche et de Ressources, Bordeaux
  - CHRU de Lille, Lille
  - CHRU de Lille, Lille (mri)
  - Hôpital Sainte-Marguerite, Marseille
  - CHU Hôpital Gui de Chaulliac, Montpellier
  - Groupe Hospitalier Broca-La Rochefoucauld, Paris
  - Clinique de L'Union, St.-Jean
  - Hôpital LA GRAVE, Toulouse
  - Chru Purpan, Toulouse
  - Clinique PASTEUR, Toulouse
- Germany (7):
  - Unversitätsklinikum Freiburg, Freiburg im Breisgau, Baden-Wurttemberg
  - Klinik fuer Psychiatrie und Psychotherapie, Charite Universitaetsmedizin Berlin, Berlin
  - Zentralinstitut fuer Seelische Gesundheit, Frankenthal
  - Klinik fuer Psychiatrie und Psychotherapie, Göttingen
  - Zentralinstitut fuer Seelische Gesundheit, Mannheim
  - Technische Universitaet Muenchen, Klinikum rechts der Isar, München
  - Universitaetsklinikum Muenster, Münster
- Spain (4):
  - Hospital del Mar, Barcelona, Barcelona
  - Hospital de la Santa Creu i Sant Pau, Barcelona, Barcelona
  - Hospital Clinico y Provincial, Barcelona, Barcelona
  - Hospital Universitario Clinico San Carlos, Madrid, Madrid

REFERENCES:
- [Derived] Pasquier F, Sadowsky C, Holstein A, Leterme Gle P, Peng Y, Jackson N, Fox NC, Ketter N, Liu E, Ryan JM; ACC-001 (QS-21) Study Team. Two Phase 2 Multiple Ascending-Dose Studies of Vanutide Cridificar (ACC-001) and QS-21 Adjuvant in Mild-to-Moderate Alzheimer's Disease. J Alzheimers Dis. 2016;51(4):1131-43. doi: 10.3233/JAD-150376. PMID 26967206
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=3134K1-200&StudyName=Study%20Evaluating%20Safety%2C%20Tolerability%2C%20And%20Immunogenicity%20Of%20ACC-001%20In%20Subjects%20With%20Mild%20To%20Moderate%20Alzheimer%27s%20Disease

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Planned duration was approximately 110 weeks (including 6 week screening period, 52 weeks of dosing, and 52 weeks of follow-up). Participants who completed the 3134K1-200-EU (B2571004) study through Week 78 had the option to exit after this time point, for continued treatment and follow-up under extension protocol 3134K1-2203-EU (B2571007).
Pre-assignment Details: The Basic Results disclose pooled data from studies NCT00479557 and NCT00498602.
Groups:
- ACC 3 µg+QS-21: Participants received 3 µg of ACC-001 and 50 µg of QS-21. Test article was given by intramuscular injection into the deltoid muscle at 0, 1, 3, 6, and 12 months.
- ACC 10 µg+QS-21: Participants received 10 µg of ACC-001 and 50 µg of QS-21. Test article was given by intramuscular injection into the deltoid muscle at 0, 1, 3, 6, and 12 months.
- ACC 30 µg+QS-21: Participants received 30 µg of ACC-001 and 50 µg of QS-21. Test article was given by intramuscular injection into the deltoid muscle at 0, 1, 3, 6, and 12 months.
- ACC 10 µg: Participants received 10 µg of ACC-001. Test article was given by intramuscular injection into the deltoid muscle at 0, 1, 3, 6, and 12 months.
- ACC 30 µg: Participants received 30 µg of ACC-001. Test article was given by intramuscular injection into the deltoid muscle at 0, 1, 3, 6, and 12 months.
- QS-21 Alone: Participants received 50 µg of QS-21. Test article was given by intramuscular injection into the deltoid muscle at 0, 1, 3, 6, and 12 months.
- Phosphate Buffered Saline: Participants received Phosphate buffered Saline (PBS). Test article was given by intramuscular injection into the deltoid muscle at 0, 1, 3, 6, and 12 months.
Period: Overall Study
Arm/Group | ACC 3 µg+QS-21 | ACC 10 µg+QS-21 | ACC 30 µg+QS-21 | ACC 10 µg | ACC 30 µg | QS-21 Alone | Phosphate Buffered Saline
Started | 36 | 61 | 40 | 35 | 12 | 44 | 17
Treated | 36 | 60 (One participant discontinued due to an AE, with an outcome of death.) | 40 | 35 | 12 | 44 | 17
Completed | 26 | 51 | 32 | 30 | 8 | 31 | 15
Not Completed | 10 | 10 | 8 | 5 | 4 | 13 | 2
Not completed — Death | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Lack of Efficacy | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 2 | 0 | 2 | 0 | 0 | 0
Not completed — Adverse Event (AE) related to Study Drug | 1 | 0 | 3 | 2 | 0 | 1 | 0
Not completed — AE not related to Study Drug | 1 | 3 | 0 | 0 | 2 | 2 | 1
Not completed — Caregiver Request | 2 | 2 | 2 | 0 | 1 | 2 | 0
Not completed — Investigator Request | 0 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Subject Request | 3 | 0 | 1 | 1 | 1 | 4 | 1
Not completed — Other | 2 | 3 | 1 | 0 | 0 | 3 | 0

BASELINE CHARACTERISTICS:
Population: 245 participants were randomized in both studies (86 participants in 3134K1-200-EU [B2571004] and 159 participants in 3134K1-2201-US [B2571005]) and included in the analysis below. One participant of the randomized participants did not receive treatment.
Groups:
- Total: Total of all reporting groups
Arm/Group | ACC 3 µg+QS-21 | ACC 10 µg+QS-21 | ACC 30 µg+QS-21 | ACC 10 µg | ACC 30 µg | QS-21 Alone | Phosphate Buffered Saline | Total
Number analyzed (Participants) | 36 | 61 | 40 | 35 | 12 | 44 | 17 | 245
Age, Continuous [Mean (Standard Deviation); unit: year] | 65.7 (7.75) | 69.3 (9.57) | 69.0 (9.27) | 71.9 (8.96) | 70.9 (9.59) | 68.8 (8.07) | 69.4 (7.82) | 69.1 (8.87)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 29 | 22 | 19 | 8 | 31 | 14 | 139
  Male | 20 | 32 | 18 | 16 | 4 | 13 | 3 | 106
Race/Ethnicity, Customized [Number; unit: number of participants]
  Asian | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
  Black or African American | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 3
  Other | 2 | 1 | 1 | 1 | 0 | 0 | 0 | 5
  White | 33 | 60 | 38 | 34 | 11 | 43 | 17 | 236
Mini-Mental State Examination (MMSE) Score [Mean (Standard Deviation); unit: score] — The MMSE was used to systematically and thoroughly assess mental status of participants. It is an 11-question measure that tests five areas of cognitive function: orientation, registration, attention and calculation, recall, and language. The total score ranges from 0 to 30. A score of 23 or lower is indicative of cognitive impairment.
  score | 21.4 (2.96) | 21.4 (3.38) | 21.0 (2.92) | 21.6 (3.16) | 21.8 (3.60) | 21.7 (3.11) | 21.2 (3.17) | 21.4 (3.13)
MMSE Stratum [Number; unit: number of participants] — The MMSE was used to systematically and thoroughly assess mental status of participants. It is an 11-question measure that tests five areas of cognitive function: orientation, registration, attention and calculation, recall, and language. The total score ranges from 0 to 30. A score of 23 or lower is indicative of cognitive impairment.
  number of participants
    High (21 - 26) | 26 | 40 | 24 | 23 | 8 | 29 | 11 | 161
    Low (16 - 20) | 10 | 21 | 16 | 12 | 4 | 15 | 6 | 84

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Treatment-emergent AEs or Serious Adverse Events (SAEs)
Description: An AE was any untoward, undesired, or unplanned clinical event in the form of signs, symptoms, disease, or laboratory or physiologic observations occurring in a person given study drug or in a sponsor's clinical study. The event did not need to be causally related to the study drug or the clinical studies. A treatment emergent AE was defined as an event that emerged during the treatment period that was absent before treatment, or worsened during the treatment period relative to the pretreatment state. An SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly.
Time Frame: approximately 110 weeks, including a 6-week screening period, 52 weeks of dosing and 54 weeks for follow-up after the last dose.
Population: The safety population included all randomized participants with documented use of at least one dose of study drug.
Measure: Number; unit: percentage of participants
Groups:
- ACC 10 µg: Participants received 10 µg of ACC. Test article was given by intramuscular injection into the deltoid muscle at 0, 1, 3, 6, and 12 months.
- ACC 30 µg: Participants received 30 µg of ACC. Test article was given by intramuscular injection into the deltoid muscle at 0, 1, 3, 6, and 12 months.
Arm/Group | ACC 3 µg+QS-21 | ACC 10 µg+QS-21 | ACC 30 µg+QS-21 | ACC 10 µg | ACC 30 µg | QS-21 Alone | Phosphate Buffered Saline
Number analyzed (Participants) | 36 | 60 | 40 | 35 | 12 | 44 | 17
percentage of participants
  Percentage of participants with AEs | 97.2 | 93.3 | 90.0 | 91.4 | 83.3 | 90.9 | 100
  Percentage of participants with SAEs | 16.7 | 18.3 | 17.5 | 14.3 | 41.7 | 11.4 | 17.6

2. Secondary Outcome: Geometric Mean Titers (GMTs) of Anti-A-beta Immunoglobulin G (IgG) Total Using an Enzyme-linked Immunosorbent Assay (ELISA) at Weeks 2, 4, 6, 8, 10, 14, 16, 24, 28, 30, 40, 50, 54, 56, 66, 78, 91, and 104
Description: The lower limit of quantification (LLOQ) was 100 U/mL and when the assay result was below LLOQ (100 U/mL), 50 U/mL was imputed for IgG.
Time Frame: Baseline, Week 2, 4, 6, 8, 10, 14, 16, 24, 28, 30, 40, 50, 54, 56, 66, 78, 91, and 104
Population: The immunogenicity population included all randomized participants with documented injection of at least one dose of study drug and at least one immunogenicity data point collected.
Measure: Geometric Mean (95% Confidence Interval); unit: U/mL
Arm/Group | ACC 3 µg+QS-21 | ACC 10 µg+QS-21 | ACC 30 µg+QS-21 | ACC 10 µg | ACC 30 µg | QS-21 Alone | Phosphate Buffered Saline
Number analyzed (Participants) | 36 | 60 | 40 | 35 | 12 | 44 | 17
U/mL
  Baseline (N: 36, 59, 40, 35, 12, 44, 17) | 50.0 [50.0 to 50.0] | 50.0 [50.0 to 50.0] | 50.0 [50.0 to 50.0] | 50.0 [50.0 to 50.0] | 50.0 [50.0 to 50.0] | 53.1 [47.1 to 59.8] | 50.0 [50.0 to 50.0]
  Week 2 (N: 35, 60, 39, 35, 12, 43, 16) | 56.6 [49.1 to 65.3] | 69.0 [57.4 to 83.0] | 86.5 [65.7 to 113.9] | 51.7 [48.3 to 55.2] | 50.0 [50.0 to 50.0] | 52.5 [47.5 to 58.1] | 50.0 [50.0 to 50.0]
  Week 4 (N: 35, 57, 38, 31, 12, 43, 16) | 53.2 [48.5 to 58.4] | 77.1 [61.9 to 96.0] | 82.8 [63.0 to 108.8] | 50.0 [50.0 to 50.0] | 50.0 [50.0 to 50.0] | 51.3 [48.7 to 53.9] | 50.0 [50.0 to 50.0]
  Week 6 (N: 36, 58, 37, 33, 12, 41, 16) | 634.8 [322.7 to 1248.5] | 1089.4 [646.0 to 1837.2] | 1343.5 [716.0 to 2521.1] | 73.4 [50.6 to 106.4] | 103.7 [38.2 to 281.4] | 50.0 [50.0 to 50.0] | 50.0 [50.0 to 50.0]
  Week 8 (N: 33, 57, 39, 33, 12, 41, 17) | 497.4 [253.5 to 976.1] | 885.2 [530.0 to 1478.7] | 1098.2 [626.9 to 1924.0] | 66.3 [48.2 to 91.1] | 99.8 [38.8 to 256.6] | 52.4 [47.6 to 57.7] | 50.0 [50.0 to 50.0]
  Week 10 (N: 34, 59, 40, 33, 12, 43, 17) | 292.3 [156.5 to 546.0] | 762.8 [468.5 to 1242.2] | 878.5 [531.3 to 1452.6] | 77.0 [48.0 to 123.3] | 94.9 [39.8 to 226.5] | 53.0 [47.1 to 59.7] | 50.0 [50.0 to 50.0]
  Week 14 (N: 33, 52, 39, 31, 11, 33, 14) | 907.5 [474.6 to 1735.6] | 2892.3 [1705.9 to 4903.8] | 3136.8 [1877.6 to 5240.7] | 89.6 [50.8 to 158.3] | 199.4 [73.7 to 539.8] | 50.0 [50.0 to 50.0] | 50.0 [50.0 to 50.0]
  Week 16 (N: 33, 59, 38, 34, 12, 41, 16) | 996.1 [487.1 to 2037.1] | 3273.2 [2083.9 to 5141.4] | 3324.7 [1959.4 to 5641.3] | 91.7 [55.2 to 152.1] | 133.9 [56.1 to 319.9] | 52.6 [47.5 to 58.1] | 50.0 [50.0 to 50.0]
  Week 24 (N: 34, 58, 37, 33, 10, 40, 16) | 547.8 [278.8 to 1076.3] | 1827.6 [1145.3 to 2916.1] | 1231.3 [712.2 to 2128.6] | 76.1 [52.1 to 111.1] | 139.1 [52.1 to 371.3] | 52.3 [47.4 to 57.4] | 50.0 [50.0 to 50.0]
  Week 28 (N: 31, 51, 33, 29, 8, 36, 16) | 2011.2 [986.9 to 4098.8] | 4299.6 [2843.8 to 6500.8] | 5407.7 [3676.0 to 7955.3] | 108.9 [61.9 to 191.8] | 334.1 [77.1 to 1448.3] | 52.4 [47.6 to 57.6] | 50.0 [50.0 to 50.0]
  Week 30 (N: 33, 56, 36, 32, 10, 38, 16) | 2028.9 [1035.8 to 3973.8] | 4316.8 [2900.2 to 6425.2] | 4713.0 [3076.0 to 7221.2] | 110.4 [64.1 to 190.0] | 234.5 [65.3 to 842.5] | 51.8 [48.2 to 55.7] | 50.0 [50.0 to 50.0]
  Week 40 (N: 32, 54, 33, 33, 9, 37, 15) | 1167.3 [609.1 to 2237.1] | 2147.2 [1407.6 to 3275.3] | 2292.9 [1436.6 to 3659.8] | 97.2 [62.4 to 151.3] | 211.0 [53.6 to 830.7] | 52.1 [47.9 to 56.7] | 50.0 [50.0 to 50.0]
  Week 50 (N: 29, 53, 33, 33, 9, 36, 16) | 937.3 [482.0 to 1822.6] | 1364.4 [911.9 to 2041.4] | 1262.3 [828.5 to 1923.2] | 80.7 [54.8 to 118.9] | 168.4 [52.4 to 541.3] | 52.8 [47.3 to 58.8] | 50.0 [50.0 to 50.0]
  Week 54 (N: 27, 51, 30, 29, 9, 29, 14) | 2031.6 [1024.2 to 4029.7] | 5744.6 [3609.1 to 9143.7] | 6677.3 [3678.7 to 12120.1] | 160.6 [69.7 to 370.2] | 491.6 [85.9 to 2812.2] | 55.0 [45.2 to 66.9] | 50.0 [50.0 to 50.0]
  Week 56 (N: 31, 52, 34, 32, 9, 34, 15) | 2635.7 [1355.5 to 5125.2] | 5906.1 [4058.8 to 8594.2] | 7642.5 [5057.9 to 11547.9] | 159.2 [74.2 to 341.8] | 463.7 [81.1 to 2650.5] | 53.4 [46.7 to 60.9] | 50.0 [50.0 to 50.0]
  Week 66 (N: 31, 54,34, 31, 9, 33, 15) | 1372.0 [717.1 to 2625.1] | 2867.4 [1835.9 to 4478.5] | 2882.2 [1793.1 to 4632.8] | 166.3 [78.8 to 350.9] | 280.0 [56.3 to 1393.9] | 63.5 [43.7 to 92.3] | 50.0 [50.0 to 50.0]
  Week 78 (N: 31, 52, 32, 32, 8, 32, 14) | 1108.4 [585.1 to 2099.4] | 1867.5 [1197.4 to 2912.5] | 1338.1 [827.3 to 2164.4] | 142.7 [71.5 to 285.1] | 256.1 [58.2 to 1128.2] | 53.6 [46.5 to 61.6] | 50.0 [50.0 to 50.0]
  Week 91 (N: 15, 9, 3, 8, 2, 6, 2) | 1824.6 [1063.2 to 3131.2] | 2497.0 [644.8 to 9670.1] | 543.0 [33.6 to 8767.8] | 76.8 [27.8 to 211.9] | 50.0 [50.0 to 50.0] | 50.0 [50.0 to 50.0] | 50.0 [50.0 to 50.0]
  Week 104 (N: 15, 9, 4, 7, 1, 6, 2) | 1326.1 [785.0 to 2240.2] | 2212.7 [406.4 to 12048.4] | 243.3 [28.8 to 2052.4] | 98.9 [30.7 to 318.3] | 50.0 [50.0 to 50.0] | 50.0 [50.0 to 50.0] | 50.0 [50.0 to 50.0]

3. Secondary Outcome: GMTs of Anti-A-beta Immunoglobulin M (IgM) Using ELISA at Weeks 2, 4, 6, 8, 10, 14, 16, 24, 28, 30, 40, 50, 54, 56, 66, 78, 91, and 104
Description: The LLOQ was 50 U/mL and when the assay result was below LLOQ (50 U/mL), 25 U/mL was imputed for IgM.
Time Frame: Baseline, Week 2, 4, 6, 8, 10, 14, 16, 24, 28, 30, 40, 50, 54, 56, 66, 78, 91, and 104
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: U/mL
Arm/Group | ACC 3 µg+QS-21 | ACC 10 µg+QS-21 | ACC 30 µg+QS-21 | ACC 10 µg | ACC 30 µg | QS-21 Alone | Phosphate Buffered Saline
Number analyzed (Participants) | 36 | 60 | 40 | 35 | 12 | 44 | 17
U/mL
  Baseline (N: 36, 59, 40, 35, 12, 44, 17) | 32.3 [24.6 to 42.4] | 38.2 [30.8 to 47.2] | 34.2 [27.7 to 42.2] | 32.9 [28.1 to 38.5] | 40.3 [27.1 to 59.9] | 30.8 [26.4 to 36.0] | 25.0 [25.0 to 25.0]
  Week 2 (N: 35, 60, 39, 35, 12,43, 16) | 85.1 [54.2 to 133.8] | 127.7 [79.5 to 205.0] | 254.5 [133.6 to 484.9] | 46.5 [32.4 to 66.7] | 76.9 [40.5 to 146.2] | 31.5 [26.6 to 37.3] | 26.5 [23.4 to 29.9]
  Week 4 (N: 35, 57, 38, 31, 12, 43, 16) | 82.3 [52.8 to 128.4] | 123.4 [75.9 to 200.7] | 276.6 [143.3 to 533.6] | 48.2 [33.2 to 70.2] | 92.0 [46.7 to 181.1] | 33.2 [28.0 to 39.3] | 27.3 [24.0 to 30.9]
  Week 6 (M: 36, 58, 37, 33, 12, 41, 16) | 626.5 [340.5 to 1152.8] | 1283.8 [742.6 to 2219.4] | 1736.6 [906.4 to 3327.1] | 72.3 [40.8 to 128.2] | 144.1 [55.9 to 371.6] | 31.1 [26.6 to 36.3] | 25.0 [25.0 to 25.0]
  Week 8 (N: 33, 57, 39, 33, 12, 41, 17) | 758.9 [388.6 to 1482.4] | 1903.8 [1097.7 to 3301.9] | 2769.5 [1407.2 to 5450.9] | 70.8 [40.8 to 123.0] | 166.4 [60.3 to 459.3] | 31.0 [26.1 to 36.8] | 26.3 [23.6 to 29.4]
  Week 10 (N: 34, 59, 40, 33, 12, 43, 17) | 595.2 [310.0 to 1143.0] | 1697.7 [980.8 to 2938.6] | 2598.1 [1382.6 to 4882.0] | 69.9 [38.3 to 127.6] | 157.1 [56.1 to 440.1] | 36.6 [28.0 to 47.9] | 27.3 [24.0 to 31.1]
  Week 14 (N: 33, 52, 39, 31, 11, 33, 14) | 770.2 [416.1 to 1425.6] | 2721.0 [1608.3 to 4603.4] | 5271.3 [2904.4 to 9567.3] | 80.8 [40.2 to 162.3] | 290.7 [71.8 to 1177.7] | 31.0 [25.5 to 37.8] | 25.0 [25.0 to 25.0]
  Week 16 (N: 33, 59, 38, 34, 12, 41, 16) | 727.3 [395.0 to 1339.0] | 3098.3 [1904.1 to 5041.2] | 5666.4 [3264.6 to 9835.3] | 93.4 [47.5 to 183.4] | 271.8 [70.5 to 1047.5] | 34.5 [27.6 to 43.0] | 25.0 [25.0 to 25.0]
  Week 24 (N: 34, 58, 37, 33, 10, 40, 16) | 461.3 [260.4 to 817.2] | 1862.5 [1137.9 to 3048.3] | 2672.4 [1553.6 to 4597.0] | 90.8 [48.1 to 171.3] | 296.2 [56.3 to 1549.6] | 30.9 [26.1 to 36.7] | 26.6 [23.3 to 30.2]
  Week 28 (N: 31, 51, 33, 29, 8, 36, 16) | 669.0 [388.0 to 1153.6] | 1915.3 [1256.2 to 2920.0] | 3593.2 [2050.4 to 6296.9] | 105.5 [50.2 to 221.6] | 590.9 [63.4 to 5511.6] | 31.3 [26.1 to 37.5] | 25.0 [25.0 to 25.0]
  Week 30 (N: 33, 56, 36, 32, 10, 38, 16) | 717.3 [432.6 to 1189.5] | 2259.4 [1524.0 to 3349.6] | 4147.2 [2423.1 to 7098.1] | 128.4 [63.1 to 261.1] | 343.3 [49.9 to 2361.4] | 37.8 [27.7 to 51.6] | 25.0 [25.0 to 25.0]
  Week 40 (N: 32, 54, 33, 33, 9, 37, 15) | 559.0 [350.7 to 891.0] | 1351.6 [885.3 to 2063.3] | 1855.9 [1074.3 to 3206.1] | 103.9 [54.2 to 199.3] | 311.9 [39.1 to 2491.7] | 34.2 [28.1 to 41.6] | 25.0 [25.0 to 25.0]
  Week 50 (N: 29, 53, 33, 33, 9, 36, 16) | 351.3 [210.2 to 587.2] | 1049.6 [701.4 to 1570.8] | 1246.4 [707.2 to 2196.7] | 84.7 [45.6 to 157.3] | 294.6 [41.2 to 2104.6] | 32.2 [27.1 to 38.3] | 25.0 [25.0 to 25.0]
  Week 54 (N: 27, 51, 30, 29, 9, 29, 14) | 477.7 [305.2 to 747.7] | 1529.1 [1045.4 to 2236.7] | 2479.5 [1373.5 to 4476.4] | 121.1 [52.1 to 281.7] | 436.9 [52.1 to 3662.2] | 36.2 [28.4 to 46.3] | 27.2 [22.7 to 32.5]
  Week 56 (N: 31, 52, 34, 32, 9, 34, 15) | 598.7 [375.1 to 955.5] | 1696.1 [1173.6 to 2451.3] | 2681.8 [1480.7 to 4857.0] | 109.8 [49.4 to 244.1] | 438.5 [51.5 to 3734.3] | 34.3 [27.2 to 43.2] | 29.5 [22.6 to 38.6]
  Week 66 (N: 31, 54, 34, 31, 9, 33, 15) | 457.6 [282.2 to 742.1] | 1422.0 [980.7 to 2061.9] | 1637.2 [961.9 to 2786.6] | 114.3 [51.6 to 253.1] | 342.1 [41.2 to 2839.9] | 36.1 [26.5 to 49.1] | 27.8 [23.8 to 32.6]
  Week 78 (N: 31, 52, 32, 32, 8, 32, 14) | 368.2 [238.4 to 568.7] | 1204.4 [815.6 to 1778.6] | 1217.7 [706.1 to 2100.1] | 107.5 [52.2 to 221.4] | 346.0 [31.2 to 3832.0] | 34.6 [27.9 to 43.0] | 28.9 [23.4 to 35.8]
  Week 91 (N: 15, 9, 3, 8, 2, 6, 2) | 391.2 [205.6 to 744.2] | 1203.4 [399.9 to 3621.9] | 679.2 [28.5 to 16208.4] | 98.9 [18.4 to 530.4] | 25.0 [25.0 to 25.0] | 28.3 [20.5 to 39.1] | 25.0 [25.0 to 25.0]
  Week 104 (N: 15, 9, 4, 7, 1, 6, 2) | 299.1 [144.2 to 620.8] | 1561.8 [438.0 to 5569.0] | 620.3 [78.8 to 4882.2] | 176.7 [26.1 to 1197.0] | 25.0 [25.0 to 25.0] | 25.0 [25.0 to 25.0] | 25.0 [25.0 to 25.0]

4. Secondary Outcome: Change From Baseline GMTs of Anti-A-beta IgG Subtypes Using ELISA at Visits Where an IgG Total Response is Measurable (at Weeks 2, 4, 6, 8, 10, 14, 16, 24, 28, 30, 40, 50, 54, 56, 66, 78, 91, and 104 if Applicable)
Description: IgG subtypes were not assessed
Time Frame: Baseline, Week 2, 4, 6, 8, 10, 14, 16, 24, 28, 30, 40, 50, 54, 56, 66, 78, 91, and 104
Groups:
- ACC 3 μg+QS-21: Participants received 3 μg of ACC-001 and 50 μg of QS-21. Test article was given by intramuscular injection into the deltoid muscle at 0, 1, 3, 6, and 12 months.
- ACC 10 μg+QS-21: Participants received 10 μg of ACC-001 and 50 μg of QS-21. Test article was given by intramuscular injection into the deltoid muscle at 0, 1, 3, 6, and 12 months.
- ACC 30 μg+QS-21: Participants received 30 μg of ACC-001 and 50 μg of QS-21. Test article was given by intramuscular injection into the deltoid muscle at 0, 1, 3, 6, and 12 months.
- ACC 10 μg: Participants received 10 μg of ACC. Test article was given by intramuscular injection into the deltoid muscle at 0, 1, 3, 6, and 12 months.
- ACC 30 μg: Participants received 30 μg of ACC. Test article was given by intramuscular injection into the deltoid muscle at 0, 1, 3, 6, and 12 months.
- QS-21 Alone: Participants received 50 μg of QS-21. Test article was given by intramuscular injection into the deltoid muscle at 0, 1, 3, 6, and 12 months.
Arm/Group | ACC 3 μg+QS-21 | ACC 10 μg+QS-21 | ACC 30 μg+QS-21 | ACC 10 μg | ACC 30 μg | QS-21 Alone | Phosphate Buffered Saline
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Approximately 110 weeks, including a 6-week screening period, 52 weeks of dosing and 54 weeks for follow-up after the last dose.
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one participant and as nonserious in another participant, or one participant may have experienced both a serious and nonserious event during the study.
Arm/Group | ACC 3 µg+QS-21 | ACC 10 µg+QS-21 | ACC 30 µg+QS-21 | ACC 10 µg | ACC 30 µg | QS-21 Alone | Phosphate Buffered Saline
Serious Adverse Events (participants affected / at risk) | 6/36 | 11/60 | 7/40 | 5/35 | 5/12 | 5/44 | 3/17
Other Adverse Events (participants affected / at risk) | 34/36 | 48/60 | 35/40 | 28/35 | 10/12 | 40/44 | 17/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ACC 3 µg+QS-21 (N=36) | ACC 10 µg+QS-21 (N=60) | ACC 30 µg+QS-21 (N=40) | ACC 10 µg (N=35) | ACC 30 µg (N=12) | QS-21 Alone (N=44) | Phosphate Buffered Saline (N=17)
Dizziness (Nervous system disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0
Syncope (Nervous system disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0
Vasogenic cerebral oedema (Nervous system disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0
Ataxia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Balance disorder (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Bradykinesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Convulsion (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Dementia Alzheimers type (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Dystonia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Embolic stroke (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Transient ischaemic attack (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Carcinoid tumour pulmonary (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Non-Hodgkins lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Uterine cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Myocardial infarction (Cardiac disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cardiac arrest (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Cyanosis (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 1 | 0 | 1 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 1
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hypotension (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Orthostatic hypotension (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Vasculitis (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Feeling cold (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Gait disturbance (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Malaise (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Oedema peripheral (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Agitation (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Confusional state (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Delusion (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hallucination (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Restlessness (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Renal failure acute (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0
Stress urinary incontinence (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Vertigo positional (Ear and labyrinth disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Intestinal obstruction (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Bile duct stone (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Clavicle fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Skin erosion (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | ACC 3 µg+QS-21 (N=36) | ACC 10 µg+QS-21 (N=60) | ACC 30 µg+QS-21 (N=40) | ACC 10 µg (N=35) | ACC 30 µg (N=12) | QS-21 Alone (N=44) | Phosphate Buffered Saline (N=17)
Injection site pain (General disorders) | 7 | 17 | 9 | 4 | 1 | 6 | 0
Fatigue (General disorders) | 5 | 7 | 4 | 1 | 0 | 5 | 1
Injection site erythema (General disorders) | 7 | 9 | 6 | 0 | 0 | 1 | 0
Injection site swelling (General disorders) | 2 | 6 | 7 | 0 | 0 | 0 | 1
Asthenia (General disorders) | 1 | 2 | 1 | 3 | 2 | 1 | 0
Oedema peripheral (General disorders) | 2 | 2 | 2 | 1 | 1 | 2 | 0
Injection site pruritus (General disorders) | 1 | 3 | 3 | 0 | 0 | 0 | 0
Gait disturbance (General disorders) | 1 | 3 | 0 | 2 | 0 | 0 | 0
Injection site induration (General disorders) | 0 | 4 | 1 | 0 | 0 | 1 | 0
Malaise (General disorders) | 2 | 1 | 1 | 0 | 2 | 0 | 0
Injection site bruising (General disorders) | 1 | 0 | 2 | 0 | 0 | 0 | 1
Injection site reaction (General disorders) | 3 | 0 | 0 | 0 | 0 | 1 | 0
Injection site warmth (General disorders) | 1 | 3 | 0 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 3 | 0 | 1 | 0 | 0 | 0
Injection site inflammation (General disorders) | 0 | 0 | 2 | 0 | 0 | 1 | 0
Irritability (General disorders) | 2 | 0 | 0 | 0 | 1 | 0 | 0
Injection site haemorrhage (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 3 | 6 | 2 | 4 | 0 | 2 | 4
Nasopharyngitis (Infections and infestations) | 4 | 6 | 1 | 2 | 0 | 4 | 1
Upper respiratory tract infection (Infections and infestations) | 3 | 3 | 5 | 3 | 1 | 1 | 1
Sinusitis (Infections and infestations) | 0 | 2 | 1 | 0 | 1 | 1 | 1
Bronchitis (Infections and infestations) | 3 | 1 | 0 | 0 | 0 | 1 | 0
Viral upper respiratory tract infection (Infections and infestations) | 1 | 2 | 0 | 1 | 1 | 0 | 0
Influenza (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 4 | 0
Oral herpes (Infections and infestations) | 0 | 2 | 0 | 1 | 0 | 0 | 1
Rhinitis (Infections and infestations) | 0 | 1 | 0 | 0 | 1 | 2 | 0
Lower respiratory tract infection (Infections and infestations) | 1 | 0 | 0 | 2 | 0 | 0 | 0
Tooth infection (Infections and infestations) | 1 | 0 | 0 | 1 | 0 | 0 | 1
Fungal skin infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 1
Furuncle (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 1
Gingivitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 1 | 0
Herpes simplex ophthalmic (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Headache (Nervous system disorders) | 3 | 14 | 4 | 2 | 0 | 8 | 1
Dizziness (Nervous system disorders) | 3 | 7 | 4 | 0 | 1 | 0 | 0
Cognitive disorder (Nervous system disorders) | 1 | 3 | 1 | 1 | 0 | 1 | 1
Somnolence (Nervous system disorders) | 1 | 2 | 0 | 0 | 1 | 1 | 1
Syncope (Nervous system disorders) | 0 | 2 | 3 | 1 | 0 | 0 | 0
Aphasia (Nervous system disorders) | 2 | 0 | 0 | 1 | 0 | 1 | 0
Dementia Alzheimers type (Nervous system disorders) | 1 | 0 | 1 | 1 | 0 | 0 | 1
Apraxia (Nervous system disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 1
Cerebral microhaemorrhage (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 1
Lethargy (Nervous system disorders) | 3 | 0 | 0 | 0 | 0 | 0 | 0
Presyncope (Nervous system disorders) | 1 | 0 | 2 | 0 | 0 | 0 | 0
Clonus (Nervous system disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0
Extrapyramidal disorder (Nervous system disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0
Sciatica (Nervous system disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0
Amnesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Memory impairment (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Mental impairment (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Migraine (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Speech disorder (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Unresponsive to stimuli (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Depression (Psychiatric disorders) | 5 | 4 | 4 | 8 | 3 | 5 | 1
Agitation (Psychiatric disorders) | 4 | 4 | 0 | 5 | 2 | 4 | 2
Anxiety (Psychiatric disorders) | 3 | 5 | 1 | 2 | 2 | 2 | 0
Confusional state (Psychiatric disorders) | 2 | 1 | 0 | 2 | 0 | 2 | 0
Abnormal dreams (Psychiatric disorders) | 3 | 0 | 1 | 1 | 0 | 0 | 0
Aggression (Psychiatric disorders) | 1 | 1 | 1 | 0 | 0 | 0 | 2
Delusion (Psychiatric disorders) | 1 | 1 | 0 | 1 | 0 | 0 | 2
Hallucination (Psychiatric disorders) | 0 | 1 | 0 | 1 | 0 | 2 | 1
Hallucination, visual (Psychiatric disorders) | 1 | 0 | 0 | 2 | 0 | 0 | 1
Paranoia (Psychiatric disorders) | 2 | 1 | 0 | 0 | 0 | 1 | 0
Delirium (Psychiatric disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 1
Depressive symptom (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 2
Disorientation (Psychiatric disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0
Hallucination, auditory (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 5 | 3 | 4 | 0 | 4 | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 5 | 4 | 1 | 0 | 2 | 2
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 3 | 2 | 2 | 0 | 4 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 | 3 | 1 | 2 | 0 | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 2 | 4 | 0 | 1 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1 | 0 | 0 | 1 | 1
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0 | 1 | 1 | 0
Bursitis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 2 | 0 | 0 | 0 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0
Torticollis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 10 | 6 | 4 | 4 | 2 | 3 | 1
Nausea (Gastrointestinal disorders) | 5 | 9 | 1 | 2 | 0 | 5 | 1
Vomiting (Gastrointestinal disorders) | 5 | 4 | 1 | 0 | 2 | 5 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 4 | 0 | 2 | 1 | 2 | 0
Constipation (Gastrointestinal disorders) | 0 | 2 | 1 | 0 | 2 | 1 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 1 | 2 | 0 | 2 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 1 | 1 | 1 | 0 | 1 | 0 | 0
Functional gastrointestinal disorder (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 3 | 3 | 3 | 4 | 1 | 9 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 1 | 3 | 1 | 0 | 3 | 1
Laceration (Injury, poisoning and procedural complications) | 1 | 3 | 1 | 0 | 1 | 1 | 0
Arthropod bite (Injury, poisoning and procedural complications) | 2 | 2 | 0 | 0 | 0 | 1 | 1
Procedural pain (Injury, poisoning and procedural complications) | 2 | 0 | 2 | 1 | 0 | 1 | 0
Excoriation (Injury, poisoning and procedural complications) | 0 | 3 | 0 | 0 | 0 | 0 | 0
Wound (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 1 | 1 | 0
Thermal burn (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 1
Skin injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Tooth fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 6 | 4 | 2 | 2 | 2 | 4 | 2
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 3 | 1 | 0 | 0 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 0 | 0 | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hypertension (Vascular disorders) | 4 | 3 | 1 | 3 | 1 | 5 | 1
Haematoma (Vascular disorders) | 0 | 1 | 1 | 0 | 0 | 4 | 1
Orthostatic hypotension (Vascular disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0
Weight decreased (Investigations) | 1 | 4 | 2 | 0 | 2 | 1 | 1
Weight increased (Investigations) | 1 | 1 | 1 | 2 | 0 | 2 | 1
Blood creatine phosphokinase increased (Investigations) | 3 | 1 | 0 | 0 | 0 | 0 | 1
Blood urea increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 1
Blood albumin decreased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Blood creatinine increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Haematocrit decreased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Haemoglobin decreased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 3 | 1 | 1 | 2 | 0 | 1 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 4 | 3 | 0 | 1 | 0 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 1 | 0 | 0 | 1
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1
Petechiae (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0
Intertrigo (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Urinary incontinence (Renal and urinary disorders) | 2 | 1 | 3 | 2 | 1 | 0 | 0
Incontinence (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1
Hydronephrosis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Renal failure (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Anaemia (Blood and lymphatic system disorders) | 1 | 1 | 1 | 1 | 0 | 2 | 1
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cataract (Eye disorders) | 0 | 3 | 1 | 1 | 1 | 0 | 0
Eye movement disorder (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 3 | 0 | 0 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1 | 1 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 2 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Breast swelling (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.